CLINICAL TRIAL: NCT06679686
Title: Effect of Digital Storytelling and Role Play on Nursing Students' Ethical Behaviours to Protect Patient Rights and Ethical Sensitivity: A Randomized Controlled Study
Brief Title: Digital Storytelling-role Play for Ethical Behaviours to Protect Patient Rights and Ethical Sensitivity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Evrim Eyikara, assistant professor, Gazi University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: GaziU-HF-ES-01
Record Dates: First submitted 2024-11-06; First posted 2024-11-07 (Actual); Last update posted 2025-05-31 (Actual); Status verified 2025-05

CONDITIONS: Analyses, Ethical; Digital Storytelling; Role Playing; Nursing Students; Ethics Education; Ethical Sensitivities; Ethical Behavior
Keywords: Digital storytelling; Role playing; Ethics Education; Ethical sensitivity; Ethical behavior
MeSH Terms: interventions — Role Playing

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Role-playing (Experimental): The role play group will make an ethical analysis of a case involving an ethical problem given to them by the researchers in the classroom environment every week and will discuss the cases using the role play method in the ethics committee to be formed after the session.
  Interventions: Other: Role Playing
- Digital storytelling (Experimental): Digital storytelling group will discuss the ethical analyses of the cases with ethical issues written by themselves outside the classroom environment. Each small group of 6-7 people will present their ethical case analyses to other group members in the classroom through digital storytelling.
  Interventions: Other: Digital Storytelling
- standard education (No Intervention): The control group will continue the standard education.

INTERVENTIONS:
Other: Role Playing — The group will analyse the instant cases given by the researchers using the role-play method.
  Arms: Role-playing
Other: Digital Storytelling — The group will analyse the ethical analysis of the cases containing ethical problems written by themselves by using digital storytelling
  Arms: Digital storytelling

SUMMARY:
This study aimed to investigate the effect of an ethics education using role-play and digital storytelling, on nursing students' ethical behaviours to protect patient's rights and ethical sensitivity.

* Is role-playing in ethics education effective in improving students' behaviours to protect patients' rights?
* Is role-playing in ethics education effective in improving students' ethical sensitivity?
* Is digital storytelling in ethics education effective in improving students' behaviours towards protecting patients' rights?
* Is digital storytelling in ethics education effective in developing students' ethical sensitivity? The researchers will compare the mean scores of the ethical behaviours toward protecting patient rights scale and ethical sensitivity scale to see whether role-playing and digital storytelling methods in ethics education have an effect on nursing students' ethical behaviours and ethical sensitivity towards protecting patient rights.
* All groups will participate in the theoretical lectures of ethics education for a total of five weeks, three hours a week.
* The theoretical lectures will consist of examination of ethics and related concepts, ethical principles, professional values in nursing, relationship between care and ethics, ethical problems and ethical approaches.
* One week after the theoretical lecture, all groups will participate in a two-week practice phase, three hours a week.
* Each group will be divided into small groups of 6-7 people.
* The Intervention I group will conduct an ethical case analysis involving an ethical problem given to them by the researchers in the classroom environment every week and will discuss the analysis using the role-play method in the ethics committee to be formed after the session.
* Intervention II group will discuss the ethical case analyses with ethical problems written by themselves by coming together outside the classroom environment.
* Each small group of 6-7 people will present their ethical case analyses to other group members in the classroom through digital storytelling.
* The control group will continue the standard education.

ELIGIBILITY:
Inclusion Criteria:

* First-time registration in the course
* Being a volunteer

Exclusion Criteria:

* Non-native speakers of the country's native language
* Previous graduation from any health-related university

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2024-11-06 (Actual); Primary Completion 2025-05-05 (Actual); Study Completion 2025-05-25 (Actual)

PRIMARY OUTCOMES:
Mean scores of ethical behaviors toward protecting patients'rights | From enrollment to the end of ethics education at 8 weeks.
  The mean score will be obtained using the ethical behaviors toward protecting patients'rights scale.
Mean scores of ethical sensitivity | From enrollment to the end of ethics education at 8 weeks.
  The mean score will be obtained using the ethical sensitivity scale.

CONTACTS AND LOCATIONS:
Locations (1):
- Gazi University Faculty of Nursing, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No